CLINICAL TRIAL: NCT05975073
Title: A Phase 1/2 Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 193 in Combination With IDE397 in Subjects With Advanced MTAP-null Solid Tumors
Brief Title: A Phase 1/2 Study of AMG 193 in Combination With IDE397 in Participants With Advanced Methylthioadenosine Phosphorylase (MTAP)-Null Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20220127
Record Dates: First submitted 2023-07-19; First posted 2023-08-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: MTAP-null Non-Small-Cell Lung Cancer; MTAP-null Solid Tumors
Keywords: Oncology; AMG 193; IDE397
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Exploration of AMG 193 Combined With IDE397 (Experimental): Participants will receive escalating doses of AMG 193 and IDE397 administered orally (PO) in cycles of 21 days.
  Interventions: Drug: AMG 193; Drug: IDE397
- Part 2: Dose Expansion of AMG 193 Combined With IDE397 (Experimental): AMG 193 and IDE397 will be administered PO in cycles of 21 days.
  Interventions: Drug: AMG 193; Drug: IDE397

INTERVENTIONS:
Drug: AMG 193 — Administered PO
Drug: IDE397 — Administered PO

SUMMARY:
The main aims of this study are to evaluate the safety and tolerability, and to determine the maximum tolerated dose (MTD) or the recommended combination dose of AMG 193 in combination with IDE397 in adult participants with metastatic or locally advanced MTAP-null solid tumors, and to evaluate the preliminary anti-tumor activity of AMG 193 in combination with IDE397 in adult participants with metastatic or locally advanced MTAP-null Non-Small-Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria

1. Evidence of homozygous loss of MTAP (null) and/or MTAP deletion.
2. Presence of advanced/metastatic solid tumor not amenable to curative treatment

   1. Part 1: MTAP-null or lost MTAP expression solid tumor for which no standard therapy exists
   2. Part 2: MTAP-null or lost MTAP expression NSCLC with progression after 1 to 2 prior lines of systemic therapy.
3. Able to swallow and retain PO administered study treatment and willing to record adherence to investigational product
4. Disease measurable as defined by RECIST v1.1
5. Adequate organ function as defined in the protocol.
6. Archived tumor tissue. Participants without archived tumor tissue available may be allowed to enroll by undergoing tumor biopsy before cycle 1 day 1 dosing.

Exclusion Criteria

1. Prior treatment with an MAT2A inhibitor or a PRMT5 inhibitor.
2. Radiologic or clinical evidence of spinal cord compression, untreated or symptomatic brain metastases or leptomeningeal disease.
3. Cardiovascular and pulmonary exclusion criteria as defined in the protocol.
4. Gastrointestinal tract disease causing the inability to take PO medication, malabsorption syndrome, requirement for IV alimentation, gastric/jejunal tube feeds, uncontrolled inflammatory gastrointestinal disease (eg, Crohn's disease, ulcerative colitis)
5. History of bowel obstruction, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of study entry.
6. Prior irradiation to > 25% of the bone marrow
7. Use of prescription medications that are known strong CYP3A4/5 inducers or strong CYP3A4/5 inhibitors within 7 days for CYP3A4/5 inhibitors, 14 days for CYP3A4/5 inducers or 5 half-lives, whichever is longer, prior to any dose of investigational medical product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) | Day 1 up to Day 21
Part 1: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 up to approximately 2.5 years
  Any clinically significant changes in vital signs, electrocardiogram (ECG), or clinical laboratory test results will be recorded as adverse events
Part 1: Number of Participants Experiencing Serious Adverse Events (SAEs) | Day 1 up to approximately 2.5 years
Part 2: Objective Response (OR) per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Day 1 up to approximately 2.5 years

SECONDARY OUTCOMES:
Part 1 and 2: Maximal Plasma Concentration (Cmax) of AMG 193 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Part 1 and 2: Cmax of IDE397 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Part 1 and 2: Time to Achieve Maximal Plasma Concentration (Tmax) of AMG 193 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Part 1 and 2: Tmax of IDE397 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Parts 1 and 2: Area Under The Curve (AUC) After Single Dose of AMG 193 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Parts 1 and 2: Area Under The Curve (AUC) After Multiple Doses of AMG 193 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Parts 1 and 2: AUC After Single Dose of IDE397 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Parts 1 and 2: AUC After Multiple Doses of IDE397 | Day 1 pre-dose up to Cycle 5 (Cycle= 21 days)
Parts 1: Overall Response per RECIST 1.1 | Day 1 up to end-of-study (EOS) (approximately 2.5 years)
Parts 1 and 2: Disease Control Rate | Day 1 up to EOS (approximately 2.5 years)
Parts 1 and 2: Time to Response (TTR) | Day 1 up to EOS (approximately 2.5 years)
Parts 1 and 2: Duration of Response (DOR) | Day 1 up to EOS (approximately 2.5 years)
Parts 1 and 2: Duration of Stable Disease | Day 1 up to EOT (approximately 6 months)
Parts 1 and 2: Progression-free Survival (PFS) | Day 1 up to EOS (approximately 2.5 years)
Parts 1 and 2: Overall Survival (OS) | Day 1 up to EOS (approximately 2.5 years)
Part 2: Number of Participants Experiencing TEAEs | Day 1 up to approximately 2.5 years
  Any clinically significant changes in vital signs, electrocardiogram (ECG), or clinical laboratory test results will be recorded as adverse events
Part 2: Number of Participants Experiencing SAEs | Day 1 up to approximately 2.5 years
Parts 1 and 2: Change From Baseline in Symmetric Dimethylation of Arginine (SDMA) in Blood | Baseline (Day 1) to EOT plus 30 days (approximately 7 months)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (27):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Community Health Network MD Anderson Cancer Center - North, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Health Partners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Astera Cancer Care, East Brunswick, New Jersey
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, Irving, Texas
- Australia (2):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Medical Centre, Clayton, Victoria
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Rigshospitalet, Copenhagen, Denmark
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Universitario Ramon y Cajal, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com